CLINICAL TRIAL: NCT01047098
Title: Effects of Taking Prenatal Vitamin-mineral Supplements During Lactation on Iron Status and Markers of Oxidation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 200816261
Record Dates: First submitted 2010-01-08; First posted 2010-01-12 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Iron Overload; Oxidative Stress; Iron-deficiency Anemia
Keywords: Lactation; Breastfeeding; Iron; Oxidative stress; Iron status and oxidative stress during lactation
MeSH Terms: conditions — Iron Overload; Anemia, Iron-Deficiency; Breast Feeding | interventions — Iron

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Iron with meals (Experimental): Prenatal vitamin without iron plus capsule containing 27 mg of iron taken with meals
  Interventions: Dietary Supplement: Iron
- Iron between meals (Experimental): Prenatal vitamin without iron plus capsule containing 27 mg of iron taken between meals
  Interventions: Dietary Supplement: Iron
- Placebo (Placebo Comparator): Prenatal vitamin without iron plus capsule containing calcium carbonate (placebo) taken between meals
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Iron — Iron as iron sulfate
  Arms: Iron with meals
Dietary Supplement: Iron — Iron as iron sulfate
  Arms: Iron between meals
Dietary Supplement: Placebo — Placebo capsule
  Arms: Placebo

SUMMARY:
Most breastfeeding women are told by their health care provider to continue taking prenatal vitamins after they give birth. A woman's requirement for iron while breastfeeding is low, yet prenatal vitamins contain a large amount of iron. The purpose of this study is to see if breastfeeding women are getting too much iron when taking prenatal vitamins.

DETAILED DESCRIPTION:
Even though iron requirements are much lower for lactating women than for pregnant or non-pregnant, non-lactating women, and iron stores during lactation are often high due to release of iron from the additional maternal erythrocytes produced during pregnancy, iron supplements are often taken by lactating women in the U.S. Many studies have shown that higher iron status is associated with higher risk of certain chronic diseases (e.g. cancer and cardiovascular diseases). The overall goal of this proposed study is to understand the potential for oxidative stress due to iron supplementation, and possible mechanisms for these effects, and to identify safe and efficacious ways to ensure adequate iron status during lactation. The specific aims are:

1. To compare markers of lipid oxidation (urinary isoprostane) and DNA damage (urinary 8-OHdG (urinary 8-hydroxy-2'-deoxyguanosine)) among 3 treatment groups: (iron given between meals (27 mg daily, in a multivitamin-mineral supplement), iron given with meals (27 mg daily, in a multivitamin-mineral supplement) and multivitamin-mineral supplement with no iron, given between meals) at the beginning and end of 3 months of treatment in 114 lactating women.
2. To compare hemoglobin and iron status (ferritin, transferrin saturation, and hepcidin) before and after treatment among the three treatment groups described above.

ELIGIBILITY:
Inclusion Criteria:

* Women less than 4 weeks postpartum
* 18 years of age or older
* Took prenatal vitamins for at least 3 months during pregnancy
* Successfully initiated breastfeeding

Exclusion Criteria:

* Anemic (Hgb < 110 g/L)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2008-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Oxidative stress | 3 month
  Isoprostane and 8-OHdG
Iron status | 3 month
  Ferritin, transferrin saturation, hepcidin

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn G Dewey, PhD, Principal Investigator — Professor
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States